CLINICAL TRIAL: NCT00938028
Title: Fecal Samples for Metabolomic and Microbiomic Studies: Effects of Preparation and Storage
Brief Title: Metabolome and Microbiomic in Fecal Samples
Acronym: MicroMet
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Harland Winter, MD, MassGeneral Hospital for Children
Other Study IDs: 2009p-000636
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Last update posted 2009-07-21 (Estimated); Status verified 2009-07

CONDITIONS: Infant
Keywords: microbiome; metabolome; stool; fecal samples; handling; toddler

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: None Retained — Stool samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Microbiome, Metabolome, Stool, Toddler: healthy infant stool samples

SUMMARY:
The purpose of this study is to evaluate the effects of storage and handling on fecal samples collected for metabolomic, proteomic and microbiomic and analysis.

DETAILED DESCRIPTION:
Background

Human fecal collection for clinical or research studies usually occurs at the residence of the subject, an environment not equipped with measures to accommodate proper preparation and storage of samples for microbiome and metabolome analysis.

Aims

To evaluate the effects of storage and handling on fecal samples collected for metabolomic, proteomic and microbiomic and analysis.

Methods

Fecal samples will be collected within several minutes of voiding from healthy infants at the time of diaper change at day-care center.

Samples will be divided into 7 tubes, and subjected to different storage temperatures, before preforming microbial analysis by DNA sequencing, and metabolome analysis by H1NMR spectroscoty.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* age 12-20 months

Ages: 12 Months to 20 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy toddlers in a day care center
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2009-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Microbiome and metabolome yield | one month

CONTACTS AND LOCATIONS:
Overall Officials: Harland Winter, MD, Principal Investigator — MGH
Locations (1):
- MassGeneral for Children, Boston, Massachusetts, United States